CLINICAL TRIAL: NCT05565508
Title: a Prospective Randomized Controlled Trial Evaluating Safe Laparoscopic Access in Patients With Previous Abdominal and Pelvic Surgery
Brief Title: Safe Laparoscopic Access in Patients With Previous Abdominal and Pelvic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Mohamed lotfy, prof. Dr, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: zuh248
Record Dates: First submitted 2022-09-27; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Laparoscopic Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- new laparoscopic access technique (Experimental): in which we used our new laparoscopic access
  Interventions: Procedure: new laparoscopic access technique for group a
- Hasson's technique (Experimental): in which we used the well-known Hasson's technique for primary laparoscopic access
  Interventions: Procedure: Hasson's technique for laparoscopic access in group b

INTERVENTIONS:
Procedure: new laparoscopic access technique for group a — new laparoscopic access technique through the epigastric region
  Other Names: new laparoscopic access technique
  Arms: new laparoscopic access technique
Procedure: Hasson's technique for laparoscopic access in group b — Hasson's technique for laparoscopic access in group b
  Arms: Hasson's technique

SUMMARY:
the study discussed the safety of new technique for primary port insertion in cases of previous abdominal and pelvic surgery

DETAILED DESCRIPTION:
the study discussed the safety of new technique for primary port insertion in cases of previous abdominal and pelvic surgery and comparing the new technique group (A) patients to already known technique called (Hasson's technique) group (B) patients

ELIGIBILITY:
Inclusion Criteria:

* Patients more than 18 year-old with history of previous abdominal and/or pelvic surgery.
* underwent laparoscopic surgery in general surgery departments in both centers from March, 2020 to july, 2022.

Exclusion Criteria:

* Patients with distended abdomen due to bowel obstruction.
* Patients with uncorrected coagulopathy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2022-07-17 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
time needed to access the peritoneal cavity | the first 15 minutes of operation
  time needed to access the peritoneal cavity
numbers of trials till the good peritoneal access achieved | the first 15 minutes of operation
  numbers of trials till the good peritoneal access achieved

SECONDARY OUTCOMES:
rate of complications | the first 15 minutes of operation
  rate of complications

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Undecided